CLINICAL TRIAL: NCT00296283
Title: An Acceptance Based Psychoeducation Intervention to Reduce Expressed Emotion in Family Members of Bipolar Patients
Brief Title: Family Workshops for Bipolar Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Miami (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20051107
Record Dates: First submitted 2006-02-23; First posted 2006-02-24 (Estimated); Last update posted 2007-05-23 (Estimated); Status verified 2007-05

CONDITIONS: Bipolar Disorder
Keywords: Relatives; Bipolar Disorder; Psychoeducation
MeSH Terms: conditions — Bipolar Disorder

INTERVENTIONS:
Behavioral: integrative behavior couples therapy

SUMMARY:
This pilot study is looking at the effects of a brief psychoeducational workshop. These one day workshops are designed to increase family members knowledge about bipolar disorder and to help with processing emotions that go along with having a relative with bipolar disorder.

ELIGIBILITY:
Inclusion Criteria:

* self-identified adult relatives of people diagnosed with bipolar disorder between ages 18 and 64; up to two persons per family can participate in the multifamily group

Exclusion Criteria:

* relative with bipolar disorder will not be involved in the workshop

Ages: 18 Years to 64 Years | Sex: All
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-08

PRIMARY OUTCOMES:
Knowledge
Anger
Attributions
Expressed Emotion

CONTACTS AND LOCATIONS:
Overall Officials: Sheri Johnson, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Coral Gables, Florida, United States